CLINICAL TRIAL: NCT04909437
Title: Efficacy of MYCOBIOTIC® In Children and Adults With Abdominal Symptoms. Double Blind, Placebo Controlled, Prospective, Cross-over Multicenter Study.
Brief Title: Efficacy of MYCOBIOTIC® in Children and Adults With Abdominal Symptoms.
Acronym: EMICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nature Science Sp. z o.o. (Industry)
Collaborators: Medical Network M. Woynarowski, J. Kierkuś Spółka jawna (MED-NET) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMICH
Record Dates: First submitted 2021-05-28; First posted 2021-06-01 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Abdominal Symptoms; Stool Culture Positive for Candida Species
Keywords: stool culture; Candida sp.; probiotic; abdominal symptoms

STUDY DESIGN:
Intervention Model Description: randomised, double blind, placebo controlled, parallel arm, cross-over
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mycobiotic group (Experimental)
  Interventions: Dietary Supplement: Mycobiotic
- Placebo group (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mycobiotic — 2 sachet/day, 21 days, oral
  Arms: Mycobiotic group
Dietary Supplement: Placebo — 2 sachet/day, 21 days, oral
  Arms: Placebo group

SUMMARY:
This is a prospective, randomised, double blind, placebo controlled, parallel arm, cross-over, multicentre study conducted in a population of children and adults with abdominal symptoms observed at outpatient primary health care centres.

ELIGIBILITY:
Inclusion criteria

1. Children and adults age >3 up to ≤ 75 years old. Boys and girls aged 3-15 years
2. Presence of abdominal symptoms
3. Informed consent for participation in the study signed by children' parents/ legal caregivers and child above 13 years old, all adults patients.

Exclusion Criteria:

1. Chronic intestinal disease, immunodeficiency or immunosuppressive treatment.
2. Chronic or acute diarrheal disease.
3. Use of laxatives or antydiarrhoeal treatment within the week before inclusion in the study.
4. Antibiotic treatment for the last four weeks before inclusion in the study.
5. Intake of probiotic products for the last two weeks before inclusion in the study
6. Known hypersensitivity to any of the ingredients in the probiotic product or the placebo (corn starch, magnesium stearate ± bacterial culture).

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
MYCOBIOTIC® influence for the intensity of abdominal pain; | Day 21+/-3; Day 42+/-3, Day 49 +/-3
  to assess if administration of MYCOBIOTIC® have influence to the intensity of the abdominal symptoms reported by parents or caregivers in questionaire- abdominal pain;
MYCOBIOTIC® influence for the intensity of stool frequency and consistency | Day 21+/-3; Day 42+/-3, Day 49 +/-3
  to assess if administration of MYCOBIOTIC® have influence to the intensity of the abdominal symptoms reported by parents or caregivers in questionaire- stool frequency and consistency
MYCOBIOTIC® influence for the intensity of abdominal distention | Day 21+/-3; Day 42+/-3, Day 49 +/-3
  to assess if administration of MYCOBIOTIC® have influence to the intensity of the abdominal symptoms reported by parents or caregivers in questionaire- abdominal distention
MYCOBIOTIC® influence for the intensity of vomiting | Day 21+/-3; Day 42+/-3, Day 49 +/-3
  to assess if administration of MYCOBIOTIC® have influence to the intensity of the abdominal symptoms reported by parents or caregivers in questionaire- vomiting
MYCOBIOTIC® influence for the intensity of abdominal bloating | Day 21+/-3; Day 42+/-3, Day 49 +/-3
  to assess if administration of MYCOBIOTIC® have influence to the intensity of the abdominal symptoms reported by parents or caregivers in questionaire- abdominal bloating

SECONDARY OUTCOMES:
Reducuction of the rate of patients with stool culture positive for Candida sp. | Day 42 +/-6
  to assess whether administration of MYCOBIOTIC® reduces the rate of patients with stool culture positive for Candida sp. in children.

CONTACTS AND LOCATIONS:
Locations (6):
- Poland (6):
  - NZOZ Promed, Kielce
  - Świętokrzyskie Centrum Pediatrii - Poradnia Gastroenterologiczna dla Dzieci, Kielce
  - Świętokrzyskie Centrum Pediatrii, Kielce
  - Prywatna Specjalistyczna Praktyka Lekarska, dr n. med. Małgorzata Sawicka-Parobczyk, Pruszków
  - Nowe Zdrowie - CK, Staszów
  - Centrum dr Ozimek, Warsaw